CLINICAL TRIAL: NCT02671058
Title: Randomized, Open Label, Crossover Study Pharmacokinetics and Bioavailability of Hydrocortisone Acetate Administered as a Suppository With the Sephure® Rectal Suppository Applicator Compared With Cortenema in Healthy Subjects
Brief Title: Pharmacokinetics and Bioavailability of Hydrocortisone Acetate Suppositories
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cristcot LLC (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CINC-2015-BA
Record Dates: First submitted 2016-01-21; First posted 2016-02-02 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: bioavailability
MeSH Terms: interventions — Hydrocortisone; hydrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cortenema (Active Comparator): Hydrocortisone retention enema (Cortenema) administered rectally as a single dose; each dose unit delivers 100 mg of hydrocortisone per 60 mL.
  Interventions: Drug: Cortenema
- Hydrocortisone acetate (Experimental): Hydrocortisone acetate suppository 90 mg administered rectally as a single dose with the Sephure Rectal Suppository Applicator
  Interventions: Drug: Hydrocortisone Acetate

INTERVENTIONS:
Drug: Cortenema — Hydrocortisone Administered as a Liquid Enema
  Arms: Cortenema
Drug: Hydrocortisone Acetate — Hydrocortisone Acetate Administered as a Suppository with the Sephure® Rectal Suppository Applicator
  Arms: Hydrocortisone acetate

SUMMARY:
This study will be an open label, single dose, randomized, 2 way (2 period) crossover study in healthy adult subjects at a single study center.

DETAILED DESCRIPTION:
This study will be an open label, single dose, randomized, 2 way (2 period) crossover study in healthy adult subjects at a single study center. Screening evaluations will occur from Day 28 to Day 2 and subjects will be confined to the clinical research unit (CRU) from Day 1 to Day 2 for each treatment period. The treatment periods will be separated by at least a 7 day washout period. Subjects meeting the study enrollment criteria will be randomly assigned to 1 of 2 sequences (AB or BA) on Day 1 of Treatment Period 1 and will receive either the reference product (A) or the treatment product (B) once during the study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 to 45 years of age, inclusive, at the time of Screening.
2. Female subjects must be:

   Of non childbearing potential (surgically sterile [hysterectomy, oophorectomy or bilateral tubal ligation] or post-menopausal >1 year with follicle stimulating hormone [FSH] > 40 U/L), or Non pregnant, non lactating females of childbearing potential who are able and willing to undertake adequate measures to prevent a pregnancy including the use of any medically acceptable forms of birth control by the subject or partner (hormonal birth control, abstinence, diaphragm with spermicide, condom with spermicide, intrauterine device, vasectomy or surgical sterilization) from Screening until the End of Study.
3. Male subjects must be able and willing to undertake adequate measures to prevent a pregnancy throughout the study including the use of any medically acceptable forms of birth control by the subject or partner (hormonal birth control, abstinence, diaphragm with spermicide, condom with spermicide, intrauterine device, vasectomy, surgical sterilization or post menopausal partner) from Screening until the End of Study.
4. Body mass index (BMI) of ≥ 18.0 and ≤ 30.0 kg/m2 at the time of Screening.
5. Subject is willing and able to provide informed consent.
6. Subject is willing and able to be confined to the CRU and adhere to the study and lifestyle restrictions.

Exclusion Criteria:

1. History of clinically significant illness or surgery as determined by the Principal Investigator or designee, within 5 years prior to the first IMP administration.
2. History or evidence of any clinically significant pathology including neurological, cardiovascular, endocrine, pulmonary, gastrointestinal, renal, hepatic, hematological, immunological, psychiatric or metabolic disorder(s) as determined by the Principal Investigator or designee.
3. Any significant rectal pathology that, in the opinion of the Principal Investigator or designee, would be a contraindication (or warning) with a hydrocortisone acetate suppository or hydrocortisone retention enema including rectal obstruction, abscess, perforation, active fungal infection(s) and/or bacterial infection(s).
4. Subject has had anal sex, cosmetic anal bleaching or perianal waxing within 30 days prior to the first IMP administration.
5. History of constipation, diarrhea or frequent bowel movements per day within 30 days prior to the first IMP administration.
6. Any clinically significant abnormality (including clinically significant laboratory test result[s]) found at Screening or febrile illness or infection within 7 days prior to Screening through Admission (Day 1 of Treatment Period 1) to the CRU.
7. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti HCV), or human immunodeficiency virus (HIV) antibody at Screening.
8. Clinically significant electrocardiogram (ECG) abnormality at Screening, as determined by the Principal Investigator or designee.
9. Positive pregnancy test (females only) at Screening or Admission (Day 1 of Treatment Periods 1 or 2) to the CRU.
10. Subject has history of alcohol abuse or of significant regular alcohol use within 1 year prior to Screening, defined as exceeding 14 units of alcohol per week, where, 1 unit = 12 ounces of beer, 5 ounces of wine or 1.5 ounces of hard liquor.
11. Positive serum alcohol test at Screening or Admission (Day 1 of Treatment Periods 1 or 2) to the CRU.
12. History of regular tobacco use or use of nicotine containing products to control tobacco use within the past 6 months prior to Screening.
13. Positive urine drug test (including amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates and phencyclidine) at Screening or Admission (Day 1 of Treatment Periods 1 or 2) to the CRU.
14. Use of over the counter (OTC) medications (including oral natural health products, vitamin and herbal supplements) within 7 days prior to the first IMP administration until the End of Study or use of prescription medication within 14 days prior to the first IMP administration until the End of Study. By exception, acetaminophen <1000 mg per day, hormonal contraception and hormonal replacement therapy are permitted.
15. Known allergy or history of hypersensitivity to hydrocortisone or any of the inert components of either of the formulations being tested.
16. Participation in another clinical study within 60 days prior to the first IMP administration. Participation is considered the last dose of IMP from another study.
17. Donation or loss of blood (> 100 mL) of either whole blood or plasma within 60 days prior to the first IMP administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
primary PK endpoints | at time 0,1, 2 and 24 hours
  Maximum plasma concentration
primary PK endpoints | at time 0,1, 2 and 24 hours
  Area under the concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Marck C Ensign, Study Chair — Executive VP Product Development

IPD SHARING:
Plan to Share IPD: No